CLINICAL TRIAL: NCT04188223
Title: Safety and Preliminary of Immunogenicity Following Recombinant Hepatitis B (Bio Farma) Vaccine in Adults & Children (Phase I)
Brief Title: Safety and Immunogenicity Following Recombinant Hepatitis B (Bio Farma) Vaccine in Adults & Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PT Bio Farma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: Hep B 0119
Record Dates: First submitted 2019-11-27; First posted 2019-12-05 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Hepatitis B
Keywords: vaccine; hepatitis b; infection; virus
MeSH Terms: conditions — Hepatitis B; Infections; Virus Diseases | interventions — Vaccines

STUDY DESIGN:
Intervention Model Description: This Study is sequential age de-escalation. To be conducted in heathy adults (18-40 years old) and followed by children (10-17 years old) )
Who Masked: Participant, Investigator
Masking Description: Double blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recombinant Hepatitis B (Bio Farma) Vaccine (Experimental): Recombinant Hepatitis B vaccine is an inactivated HbsAg produced in yeast cells (Hansenula polymorpha) using recombinant DNA technology. It is a whitish liquid produced by culture genetically engineered yeast cell which carry the relevant gene of the HbsAg and purified and inactivated by several physicochemical steps such as ultracentrifugation, column chromatography and formaldehyde treatment.
  Interventions: Biological: Recombinant Hepatitis B (Bio Farma) Vaccine
- Control Product: Recombinant Hepatitis B (Bio Farma) Vaccine® (Active Comparator): Registered Recombinant Hepatitis B vaccine is an inactivated HbsAg produced in yeast cells (Hansenula polymorpha) using recombinant DNA technology. It is a whitish liquid produced by culture genetically engineered yeast cell which carry the relevant gene of the HbsAg and purified and inactivated by several physicochemical steps such as ultracentrifugation, column chromatography and formaldehyde treatment.
  Interventions: Biological: Recombinant Hepatitis B (Bio Farma) Vaccine®

INTERVENTIONS:
Biological: Recombinant Hepatitis B (Bio Farma) Vaccine — Recombinant Hepatitis B vaccine produced by Bio Farma
  Arms: Recombinant Hepatitis B (Bio Farma) Vaccine
Biological: Recombinant Hepatitis B (Bio Farma) Vaccine® — Registered Recombinant Hepatitis B vaccine produced by Bio Farma
  Arms: Control Product: Recombinant Hepatitis B (Bio Farma) Vaccine®

SUMMARY:
This trial is an experimental, randomized, double blind, prospective intervention study

Approximately 100 subjects will be enrolled in this trial, divided into 2 arms, as follow:

For adult (18-40 years old)

DETAILED DESCRIPTION:
Each study age group/arm will be divided into two groups of treatment. One group will receive investigational product and one other group will receive active comparator. This Study is sequential age de-escalation. To be conducted in heathy adults (18-40 years old) and followed by children (10-17 years old) ). Before the study started, the subjects will be assessed for anti HBs Antibody. For subjects with anti-HBs not protective (< 10mIU/mL) before immunization, additional 2 doses will be required with 1 month interval.

ELIGIBILITY:
Inclusion Criteria:

Adult

1. Healthy individu as determined by clinical judgment, including a medical history, physical exam, rontgen thorax and laboratory results, which confirms the absence of a current or past disease state considered significant by the investigator.
2. Subjects have been informed properly regarding the study and signed the informed consent form
3. Subjects will commit to comply with the instructions of the investigator and the schedule of the trial

Children:

1. Healthy individu as determined by clinical judgment, including a medical history, physical exam and rontgen thorax which confirms the absence of a current or past disease state considered significant by the investigator.
2. Subjects/parents/guardian(s) have been informed properly regarding the study and signed the informed consent form and
3. Subject/parents/guardian(s) will commit to comply with the instructions of the investigator and the schedule of the trial.

Exclusion Criteria:

1. Subject concomitantly enrolled or scheduled to be enrolled in another trial
2. Any direct relatives relationship with the study team.
3. Evolving mild, moderate or severe illness, especially infectious diseases or fever (axillary temperature ³ 37.5°C) within the 48 hours preceding enrollment.
4. Known history of allergy to any component of the vaccines (based on anamnesis)
5. Known history of immunodeficiency disorder (HIV infection, leukemia, lymphoma, or malignancy)
6. History of uncontrolled coagulopathy or blood disorders contraindicating for phlebotomy.
7. Subject who has received in the previous 4 weeks a treatment likely to alter the immune response (intravenous immunoglobulins, blood-derived products, or corticosteroid therapy and other immunosuppresant).
8. Any abnormality or chronic disease which according to the investigator might interfere with the assessment of the trial objectives.
9. Pregnancy or planning a pregnancy within the next 3 months & lactation. (for Adults)
10. Subject already immunized with any vaccine within 4 weeks prior and expects to receive other vaccines within 4 weeks following immunization.
11. HbsAg positive
12. Subjects with known history of Hepatitis B infection.
13. Subjects who have received Hepatitis B vaccination which proven by vaccination records.
14. Subject planning to move from the study area before the end of study period.

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2020-07-16 (Actual); Study Completion 2020-07-16 (Actual)

PRIMARY OUTCOMES:
Number of subjects with Immediate reaction | 3 months
  Number of subjects with at least one immediate reaction (local reaction or systemic event) within 30 minutes after one dose or three doses of Hepatits B vaccination
percentage of subjects with Immediate reaction | 3 months
  Percentage of subjects with at least one immediate reaction (local reaction or systemic event) within 30 minutes after one dose or three doses of Hepatits B vaccination

SECONDARY OUTCOMES:
Number of subjects with Adverse Events from 1 day to 28 days after vaccination | 3 months
  Number of subjects with at least one of these adverse events, solicited or not, within 24 h, 48h, 72h and 28 days after each dose vaccination
Percentage of subjects with Adverse Events from 1 day to 28 days after vaccination | 3 months
  Percentage of subjects with at least one of these adverse events, solicited or not, within 24 h, 48h, 72h and 28 days after each dose vaccination
Number of subjects with Serious Adverse Events from 1 day to 28 days after vaccination | 3 Months
  Number of subjects with serious adverse event from inclusion until 28 day after each dose vaccination.
Percentage of subjects with serious Adverse Events from 1 day to 28 days after vaccination | 3 Months
  Percentage of subjects with serious adverse event from inclusion until 28 day after each dose vaccination.
Number of Lab Deviation for adults subjects in 7 days of immunization | 7 Days After 1st Vaccination
  Number of deviation from routine biochemical (SGOT, SGPT, Ureum, Creatinine) and Hematological (Hb, Hct, Dif, Leucocyte count, Total Leucocyte, total Eryhrocyte, total Thrombocyte) laboratory evaluation that probably related to the vaccination (adults subject).
Safety Comparison between each intervention group | 3 months
  incidence of any adverse event, compared between two intervention arms
Protectivity of Hepatitis B vaccine (number of subject with protective anti HbsAg) | 3 months
  Number of subjects with anti-HbsAg more than 10mIU/ml, 28 days after 1 dose or three doses of vaccination.
Protectivity of Hepatitis B vaccine (4 times increasing antibody) | 3 months
  - Number and percentage of subjects with more than 4 folds increasing antibody
Protectivity of Hepatitis B vaccine (Geometic Mean Titers) | 3 months
  - Geometric Mean Titers (GMT) following immunization
Anti-HBs description between groups | 3 months
  Number of subjects with protective Anti-HBs value, compared between intervention groups after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Kusnandi Rusmil, Professor, Principal Investigator — Padjadjaran University
Locations (1):
- Hasan Sadikin Hospital, Bandung, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No